CLINICAL TRIAL: NCT02521155
Title: "Safeguard Your Smile" an Oral Health Literacy Intervention Promoting Positive Oral Hygiene Self-care Behavior Among Punjabi Immigrants: A Randomized Controlled Trial
Brief Title: "Safeguard Your Smile" an Oral Health Literacy Intervention Promoting Positive Oral Hygiene Self-care Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Louise Potvin, Canada Research Chair (950-228295), Institut de recherche en Santé Publique and the Centre de Recherche Léa-Roback, School of Public Health, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-071-CERES-D
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2015-09

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Oral health literacy intervention; oral hygiene behavior
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Safeguard Your Smile an oral health literacy intervention.
  Interventions: Behavioral: Safeguard Your Smile an oral health literacy intervention
- Control group (No Intervention): No intervention, only a conventional pamphlet will be given.

INTERVENTIONS:
Behavioral: Safeguard Your Smile an oral health literacy intervention — Safeguard Your Smile intervention will consist of following five components:
  i) Reviewing photonovel (educational booklet) with participants to help them understand adequate oral hygiene self-care behavior. ii) Demonstrating adequate tooth brushing, flossing and tongue cleaning (frequency, duration and technique) on dentoform iii) Helping participants to make a concrete plan (specifying when where and how will they perform oral hygiene self-care behavior and a coping plan). Also, to identify a prompt/cue that would act as a reminder. iv) Assigning a task to participants to daily check-mark their behavioral progress on a calendar provided in the photonovel for the next three months. v) Follow up by making three phone calls to each participant of the intervention group once a month.
  Arms: Intervention group

SUMMARY:
The purpose of the investigators' study is to assess effectiveness of community based oral health literacy intervention promoting positive oral hygiene self-care behavior among Montreal's Punjabi immigrants.

DETAILED DESCRIPTION:
There will be 140 participants in this study who will be randomly allocated into either intervention group (70) or control group (70).The intervention group will receive one hour long "Safeguard Your Smile" intervention and control group will receive no intervention and only a conventional pamphlet. Data will be collected at baseline and after 3 months using three research instruments. i) Oral hygiene self-care knowledge and oral hygiene self-care behavior will be assessed using self administered questionnaire. ii) Using Loe and Sillness indices, plaque and gingival index scores will be measured. iii) And oral health literacy of participants will be measured with the TS-REALD tool.The data analysis will include descriptive statistics and frequency tables will be provided for both baseline and endpoint data of the both groups. Continuous variables will be summarized with mean, standard deviation and range and for the categorical variables; frequency counts and percentage of subjects within each category will be provided. An array of data analysis including t-test, correlations and logistic regression will be performed assessing effectiveness of the Safeguard Your Smile intervention.

ELIGIBILITY:
Inclusion Criteria:

* Punjabi immigrants who are Montreal residents
* Be in good general health
* Will give written informed consent

Exclusion Criteria:

* Non permanent residents e.g. refugees
* Presence of orthodontic appliances
* Having any disease of soft/ hard oral tissues e.g. advanced periodontitis
* Having any systemic disease e.g. diabetes
* On certain medications such as phenytoin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Oral hygiene self-care knowledge using a self administered questionnaire | Three months
  Using a self administered questionnaire
Oral hygiene self-care behavior using a self administered questionnaire | Three months
  Using a self administered questionnaire
Gingival index | Three months
  Loe and Sillness gingival index scores to assess gingivitis, score 0=no gingival inflammation, 1=mild inflammation-slight change in colour of gingiva, 2=moderate inflammation-moderate glazing, redness, edema and hypertrophy, tendency to bleed, score 3=severe inflammation, marked redness and hypertrophy, tendency to spontaneous bleeding.
Dental plaque index | Three months
  Loe and Sillness plaque index on the six Ramfjord teeth (16, 12, 24, 36, 32, 44 on proximal, buccal and lingual sides). Score 0= no dental plaque seen in the gingival area; score 1= dental plaque present on the free gingival margin; score 2= moderate accumulation of dental plaque at the gingival margin seen by naked eye and score 3= abundant dental plaque in the gingival margin.

SECONDARY OUTCOMES:
Oral health literacy measured using TS-REALD (Two Stage Rapid Estimate of Adult Literacy in Dentistry) | Three months
  Participant's oral health literacy levels will be measured using validated oral health literacy measurement instrument i.e. TS-REALD (Two Stage Rapid Estimate of Adult Literacy in Dentistry). TS-REALD is a word recognition routing test in which participants are asked to read a list of 5 dental words aloud and one point is given for the correct answer. This first stage of the test categorizes the participants depending on their scores into three groups of stage 2 for further testing: i) low literacy stage-2 (4 words test); ii) average literacy stage-2 (6 words test); and high literacy stage-2 ( 3 words test).The score from routing test is added to stage-2 score and this is called raw score. This raw score is translated into a scaled score by using the scaled score translational table that had been derived using psychometric testing. Specific cut offs for high and low oral health literacy are determined using the mean and the standard deviation of the scaled scores.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Potvin, BA MSc. PhD, Study Director — Université de Montréal; Daniel P. Kandelman, DrCD DMD MPH, Study Director — Université de Montréal; Navdeep Kaur, BDS MSc., Principal Investigator — Université de Montréal
Locations (1):
- Faculty of Dental medicine, Montreal, Quebec, Canada